CLINICAL TRIAL: NCT07120269
Title: Predictive Markers of the Course of Covid-19 Based on Biomarker Serum Amyloid A (SAA) and Genetic Markers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomayer University Hospital (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Martina Koziar Vašáková, Head of the Department of Respiratory Medicine, Thomayer University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2511/21 + 4687/21
Record Dates: First submitted 2025-08-01; First posted 2025-08-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: COVID-19; Serum Amyloid A; Predictive markers
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control Group (Experimental): Individuals without prior SARS-CoV-2 infection and with a negative RT-PCR result
  Interventions: Diagnostic Test: Nasal swab to collect material for RT-PCR SAA evaluation
- asymptomatic (Experimental): Individuals with an asymptomatic course of SARS-CoV-2 infection
  Interventions: Diagnostic Test: Nasal swab to collect material for RT-PCR SAA evaluation
- mild and moderate (Experimental): Individuals with a moderate course of SARS-CoV-2 infection (without hospitalization)
  Interventions: Diagnostic Test: Nasal swab to collect material for RT-PCR SAA evaluation
- Severe (Experimental): Individuals with a severe course of SARS-CoV-2 infection (requiring hospitalization)
  Interventions: Diagnostic Test: Nasal swab to collect material for RT-PCR SAA evaluation
- Severe ICU (Experimental): Individuals with a severe course of SARS-CoV-2 infection (requiring hospitalization in intensive care units)
  Interventions: Diagnostic Test: Nasal swab to collect material for RT-PCR SAA evaluation
- Severe below 40 (Experimental): Individuals from study arms 4 and 5 aged below 40 years.
  Interventions: Diagnostic Test: Nasal swab to collect material for RT-PCR SAA evaluation

INTERVENTIONS:
Diagnostic Test: Nasal swab to collect material for RT-PCR SAA evaluation — Nasal swab for parallel identification of SARS-Cov2 and SAA expression

SUMMARY:
This study focuses on identifying genetic and biochemical markers (biomarkers) that could help predict the course of COVID-19. The investigators aim to analyze samples taken from the nasopharynx (nose and throat), saliva, and blood of patients with acute respiratory tract infections who come to the Outpatient Clinic of the Department of Respiratory Diseases at the Thomayer University Hospital.

The main objectives include measuring the expression of the SAA1 gene (using quantitative RT-PCR) and conducting broader gene expression analysis (using RNA sequencing) in nasopharyngeal cells. At the same time, the investigators will examine the patients' DNA to identify rare genetic variants or common polymorphisms that may influence their immune response to the virus.

The goal is to relate the values of SAA expression with clinical and radiological status and outcome of the patients. The investigators hypothesize, that SAA may predict the severity of the disease, need for hospitalizastion and outcome of the patients.

DETAILED DESCRIPTION:
This cross-sectional study evaluated nasal SAA1 expression as a biomarker for early detection and severity assessment of respiratory tract infections, particularly in COVID-19 patients. A total of 369 participants presenting with infectious or non-infectious respiratory symptoms to the outpatient clinic were prospectively recruited between March 6, 2021, and June 26, 2023.

Each patient underwent a single nasopharyngeal swab, which was used both for RT-qPCR testing of SARS-CoV-2 RNA and for SAA1 expression analysis, ensuring methodological consistency and direct comparability of results. Additionally, all participants underwent a chest X-ray, a comprehensive clinical examination, and routine blood and biochemistry testing.

RNA Extraction and SAA1 mRNA Quantification:

Nasal swabs were collected and stored under RNase-free conditions for RNA extraction. The relative expression of SAA1 was determined using real-time quantitative polymerase chain reaction (RT-qPCR).

ELIGIBILITY:
Inclusion Criteria:

* The patients coming to the outpatient clinic and emergency room of the Department of Respiratory Diseases in Thomayer Hospital with symptoms of acute respiratory infection

Exclusion Criteria:

* Inability to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The ability of SAA expression to predict clinical picture and outcome of the disease | 14 days
  Levels of expression of SAA are related to the risk of hospitalization for COVID-19
The ability of SAA expression to predict risk of death for COVID-19 | 3 months
  Levels of expression of SAA are related to the risk of death

CONTACTS AND LOCATIONS:
Locations (1):
- Thomayer University Hospital, Department of Respiratory Medicine, Prague, Czechia